CLINICAL TRIAL: NCT04075071
Title: A Pilot Study of Teacher-Child Interaction Training - Universal in Head Start
Acronym: TCIT-U
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Intervention and and final data collection point was not completed due to coronavirus school closures in March 2020.
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: PNC Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-016084; IRB 19-016084 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2019-08-13; First posted 2019-08-30 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Child Behavior; Child Development; Child Behavior Problem
Keywords: Teacher-Child Interaction Training; teacher-child relationships; child behavior; child social-emotional skills; preschool; teaching self-efficacy; teacher behavior
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCIT-U (Experimental): Four teachers from two Head Start classrooms will be assigned to Teacher-Child Interaction Training - Universal (TCIT-U). TCIT-U occurs in two phases (6 weeks per phase): Child-Directed Interaction (CDI; focusing on relationship building) and Teacher-Directed Interaction (TDI; focusing on managing behavior problems). The TCIT-U Trainer (a licensed clinical child psychologist) will provide teachers with group didactic sessions (6 hours per phase) and individualized live coaching in their classrooms (20 minutes, once per week). Strategies include the use of PRIDE skills (Praise, Reflection, Imitation, Behavior Description, and Enthusiasm) or specific verbalizations that promote warm, responsive interactions, as well as classroom-appropriate behavior modification strategies which include using effective commands, prompts, natural consequences, differential social attention, and a modified time-out appropriate for use in a classroom.
  Interventions: Behavioral: Teacher-Child Interaction Training - Universal
- Usual Care (No Intervention): Four teachers from 2 PreK Counts classrooms will be assigned to the Usual Care (UC) group. They will continue their existing behavioral management strategies and techniques. Teachers will report on specific training in and use of other behavior management and social-emotional learning programs at baseline. At the conclusion of the study, UC teachers and staff will be offered didactic training in TCIT-U principles and strategies.

INTERVENTIONS:
Behavioral: Teacher-Child Interaction Training - Universal — Teacher-Child Interaction Training - Universal (TCIT-U) is an empirically-supported classroom-based intervention designed to strengthen teacher-child relationships, reduce and prevent child behavior problems, and promote social-emotional skills. TCIT-U is based in behavioral and attachment principles and was developed as a modification of Parent-Child Interaction Therapy (PCIT), an evidence-based treatment with well-established support for decreasing disruptive child behaviors and parental stress with children ages two to seven years old. In TCIT-U, teachers of children, preschool through second grade, are taught and coached in skills to manage challenging classroom behaviors and improve the quality of relationships. TCIT-U is delivered to teachers through group didactic training and live individualized coaching.
  Arms: TCIT-U

SUMMARY:
This pilot study aims to implement and evaluate Teacher-Child Interaction Training - Universal (TCIT-U), an empirically-supported classroom-based intervention aimed at improving child behavior and social-emotional skills through strengthening teacher-child relationships at a preschool that serves children from socially and economically disadvantaged backgrounds who are at risk for behavioral health difficulties. The main objectives are to (a) examine TCIT-U's effects on teacher behavior, teachers' sense of efficacy, and child behavior problems and social-emotional skills compared to usual care (UC) and (b) explore the feasibility and acceptability of implementing TCIT-U at a diverse urban preschool.

DETAILED DESCRIPTION:
Disruptive behaviors and social-emotional skill deficits are common problems in early education settings and contribute to the high rates of preschool suspensions and expulsions. While teachers serve a critical role in children's behavioral health, they often lack evidence-based training in strategies that could improve child behavior and promote social-emotional skills. The goal of this project is to implement and evaluate Teacher-Child Interaction Training - Universal (TCIT-U), an empirically-supported classroom-based intervention aimed at improving child behavior and social-emotional skills through strengthening teacher-child relationships at a preschool that serves children from socially and economically disadvantaged backgrounds who are at risk for behavioral health difficulties.

The main objectives are to (a) examine TCIT-U's effects on teacher behavior, teachers' sense of efficacy, and child behavior problems and social-emotional skills compared to usual care (UC) and (b) explore the feasibility and acceptability of implementing TCIT-U at a diverse urban preschool.

This pilot study is a nonrandomized clinical trial comparing TCIT-U to a UC control group at urban preschool. Teachers in the intervention group will participate in TCIT-U. TCIT-U and UC teachers will complete measures at baseline, post-intervention, and end-of-the-school-year follow-up. All teachers will be observed for their TCIT-U skill use at baseline, mid-intervention, post-intervention, and follow-up. Qualitative interviews will be conducted with educational staff at follow-up to examine feasibility and acceptability data.

Participants will be eight teachers and approximately 80 children from four preschool classrooms in Philadelphia. Educational staff will also be invited to participate in qualitative interviews. Staff must speak English to participate. There is no exclusion criteria for children.

Four teachers from two Head Start classrooms will participate in TCIT-U. TCIT-U is an empirically-supported intervention aimed at strengthening teacher-child relationships and improving child behavior and social-emotional skills. TCIT-U includes group didactic and individualized coaching sessions. Four teachers from two other classrooms will serve as the UC control group.

Teacher behavior will be coded during live classroom observations. Teacher-reported questionnaires will measure teachers' sense of efficacy and child behavior and social-emotional skills. Qualitative interviews and satisfaction surveys will explore the feasibility and acceptability of implementing TCIT-U. Fidelity checklists will be completed by the TCIT-U Trainer and expert consultants to document intervention fidelity.

ELIGIBILITY:
Teachers' Inclusion Criteria:

* Serve as a head, co-, and/or assistant teacher in a Head Start or PreK Counts classroom at the participating early childhood education center.
* Speak and read English proficiently.
* Provide written informed consent.

Teachers' Exclusion Criteria: Do not speak and read English proficiently.

Children's Inclusion Criteria:

* Enrolled in one of the participating Head Start or PreK Counts classrooms prior to baseline evaluations.
* Aged 3 through 5 years old.
* Provided an informational letter about the study to their parents.

Children's Exclusion Criteria: There are no exclusion criteria for children.

Educational Staff's Inclusion Criteria (qualitative interviews):

* Participated in or observed TCIT-U training and/or serve as a classroom-based (e.g., assistant, behavioral specialist) or administrative (e.g., center director) staff for the classrooms participating in TCIT-U.
* Speak and read English proficiently.
* Provide written informed consent.

Educational Staff's Exclusion Criteria (qualitative interviews): Do not speak and read English proficiently.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Changes in Teacher-Child Interaction Coding System (TCICS) | Week 1, Week 6-8, Week 12, and Month 10
  Teachers' use and maintenance of skills taught in TCIT-U will be measured using the Teacher-Child Interaction Coding System (TCICS; Budd & Stern, 2019), an observational coding system that has been used in prior TCIT-U projects and was adapted from the coding system used in PCIT (Dyadic Parent-Child Interaction Coding System, 4th edition; Eyberg, Chase, Fernandez, & Nelson, 2014). RAs, blind to study condition, will tally teachers' verbalizations (Labeled Praises, Reflections, Descriptions, Questions, Commands, and Negative Talk) during 5-minute intervals which will be conducted three times at each data collection time-point (baseline, mid-intervention, post-intervention, and follow-up).

SECONDARY OUTCOMES:
Teachers' Sense of Efficacy Scale (TSES) | Week 1, Week 12, and Month 10
  Teachers' beliefs in their capability of influencing factors related to academic instruction and student behavior will be assessed using the Teachers' Sense of Efficacy Scale (TSES; Tschannen-Moran & Woolfolk Hoy, 2001). Teachers will rate their perceived efficacy in three areas (Student Engagement, Instructional Practices, and Classroom Management) at baseline, post-intervention, and follow-up. The rating is based on a scale of 1 (nothing), to 9 (a great deal).
Devereux Early Childhood Assessment for Preschoolers, 2nd Edition (DECA-P2) | Week 1, Week 12, and Month 10
  Child behavior problems (e.g., noncompliance, aggression) and social-emotional skills (e.g., self-regulation) will be assessed using the Devereux Early Childhood Assessment for Preschoolers, Second Edition (DECA-P2; LeBuffe & Naglieri, 2012). The DECA-P2 is a 38-item standardized, strengths-based behavior rating scale that yields a Total Protective Factors scale (Initiative, Self-Regulation, Attachment/Relationships) and a Behavioral Concerns scale. Teachers will rate the frequency of children's behavior at baseline, post-intervention, and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca M Kanine, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No